CLINICAL TRIAL: NCT06586788
Title: Validation of Indiana's Early Neurodevelopmental Evaluation Hub Program
Brief Title: Validation of Indiana's Early Evaluation Hub System
Acronym: EAER21
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Purdue University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Rebecca McNally Keehn, Assistant Professor of Pediatrics, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1806262614; R21MH121747 (NIH)
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Results first posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Autism
Keywords: primary care; biomarkers; eye-tracking; diagnosis
MeSH Terms: conditions — Autistic Disorder; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Children Undergoing Developmental Evaluation (Experimental): Participating EE Hubs referred a prospective, consecutive sample of children who received an EE Hub evaluation. Next, the study team traveled to the EE Hub to conduct a follow-up gold-standard autism diagnostic assessment (reference standard diagnosis) and eye-tracking biomarker battery (index test; Aim 2) within 16 weeks of EE Hub evaluation. Reference standard diagnosis was made by a licensed clinical psychologist with expertise in autism diagnosis based upon a research evaluation including the Autism Diagnostic Observation Schedule, Second Edition (ADOS-2), Vineland Adaptive Behaviors Scale, Third Edition (VABS-3), Mullen Scales of Early Learning (MSEL), and a caregiver interview to assess for DSM-5 autism criteria. Children also completed a short (< 15min) eye-tracking activity where the children view a series of different images/videos while the children's eye movements and pupil diameter was measured.
  Interventions: Diagnostic Test: Eyelink Portable Duo; Diagnostic Test: Integrated PCP Diagnosis and Eye-tracking Biomarker

INTERVENTIONS:
Diagnostic Test: Eyelink Portable Duo — Eye-tracking data will be collected using a commercially-available remote eye-tracking system (Eyelink Portable Duo). Eye movements and pupil diameter will be collected while participants view a series of developmentally appropriate pictures and movies. The eye-tracker consists of two cameras; one that monitors eye movements and a second scene camera that monitors head movements, which permits eye tracking to take place without any equipment touching the child. Children will be asked to sit in highchair or on a caregiver's lap and will face a computer monitor. After a sticker is applied to the child's forehead and brief eye-movement calibration completed, next visual stimuli (i.e., pictures and videos) will be presented on a laptop computer monitor that is placed at approximately 60-80cm from the child. The eye tracking portion of the visit will last approximately 15 minutes or until the child is no longer able to attend to pictures/videos.
Diagnostic Test: Integrated PCP Diagnosis and Eye-tracking Biomarker — A Classification and Regression Tree (CART) Analysis, based on recursive partitioning, was used to determine which combination of variables (EE Hub PCP diagnosis, diagnostic certainty, composite biomarker, and biomarker frequency [sum of all individual biomarkers (0-6) that exceeded the 95% specificity threshold for each child]) best predicted reference standard autism diagnosis.

SUMMARY:
The investigators' objective is to test an innovative method of autism diagnosis that integrates clinical evaluation and assessment of biobehavioral markers in a large high-risk community-referral sample of children in the primary care setting.

DETAILED DESCRIPTION:
Determine whether eye-tracking biomarkers can reliably differentiate young children with and without autism in a community referred sample. The study will use a non-invasive remote eye-tracking system (Eyelink Portable Duo) to acquire a short series (less than 15 mins) of eye-tracking measures (e.g., looking time, pupil diameter, oculomotor dynamics), which may be associated with autism in young children. Differences in metrics between children with and without autism will be compared to validate potential eye-tracking biomarkers.

Determine whether a combination of clinical (i.e., EE Hub PCP measures) and eye-tracking biomarkers can be used to accurately predict autism diagnostic outcome in a sample of young children evaluated for autism in the primary care setting.

ELIGIBILITY:
Inclusion Criteria:

Young children ages 14-48 months seen at an EE hub and referred for a comprehensive autism evaluation.

Children must have English-speaking caregivers. Children must have a legal guardian that is able to provide consent.

Exclusion Criteria:

Child is younger than 14 months or older than 48 months. Child's caregiver(s) is/are not English-speaking.

Ages: 14 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 154 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca McNally-Keehn, PhD, HSPP, Principal Investigator — IU School of Medicine; Brandon Keehn, PhD, Principal Investigator — Purdue University
Locations (7):
- United States (7):
  - Community Health Network, Anderson, Indiana
  - Margaret Mary Health Pediatrics, Batesville, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - Meridian Health Pediatrics, Muncie, Indiana
  - Deaconess Riley Children's Specialty Center, Newburgh, Indiana
  - Primary Care Partners of South Bend, South Bend, Indiana
  - Lutheran Health Physicians Pediatric Healthcare, Warsaw, Indiana

IPD SHARING:
Plan to Share IPD: Yes
Data from this study is submitted to the National Institute of Mental Health Data Archive (NDA). NDA is a data repository run by the National Institute of Mental Health (NIMH) that allows researchers studying autism and other conditions to collect and share deidentified information with each other. A data repository is a large database where information from many studies is stored and managed.
  During and after the study, the researchers will send deidentified information to NDA. Other researchers nationwide can then file an application with the NIMH to obtain access deidentified study data for research purposes.
Time Frame: Investigators will follow NIMH NDAR policies for submission of data.
Access Criteria: Investigators will follow NIMH NDAR policies for submission of data. Other researchers nationwide can file an application with the NIMH to obtain access deidentified study data for research purposes.
URL: https://nda.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seven EE Hubs set within primary care practices referred children, ages 14-48 months evaluated for autism in the community primary care setting, to the study between June 2019 and August 2022. To be included, children were age 14-48 months at time of EE Hub evaluation and had an English-speaking primary caregiver/guardian. Participating EE Hubs referred a prospective, consecutive sample of children who received an EE Hub evaluation.
Groups:
- Children Undergoing Developmental Evaluation: Eyelink Portable Duo: Eye-tracking data will be collected using a commercially-available remote eye-tracking system (Eyelink Portable Duo). Eye movements and pupil diameter will be collected while participants view a series of developmentally appropriate pictures and movies. Children will be asked to sit in highchair or on a caregiver's lap and will face a computer monitor. After a sticker is applied to the child's forehead and brief eye-movement calibration completed, next visual stimuli (i.e., pictures and videos) will be presented on a laptop computer monitor that is placed at approximately 60-80cm from the child. The eye tracking portion of the visit will last approximately 15 minutes or until the child is no longer able to attend to pictures/videos.
  Integrated PCP Diagnosis and Eye-tracking Biomarker: A Classification and Regression Tree (CART) Analysis, based on recursive partitioning, was used to determine diagnostic outcome based on PCP diagnosis, diagnostic certainty, and biomarker measures.
Period: Overall Study
Arm/Group | Children Undergoing Developmental Evaluation
Started | 154
Completed | 146
Not Completed | 8
Not completed — Eye-tracking calibration / validation could not be completed with eight children | 8

BASELINE CHARACTERISTICS:
Population: Included participants
Groups:
- Children Undergoing Developmental Evaluation: Participating EE Hubs referred a prospective, consecutive sample of children who received an EE Hub evaluation. Reference standard diagnosis was made by a licensed clinical psychologist with expertise in autism diagnosis based upon a research evaluation including the Autism Diagnostic Observation Schedule, Second Edition (ADOS-2), Vineland Adaptive Behaviors Scale, Third Edition (VABS-3), Mullen Scales of Early Learning (MSEL), and a caregiver interview to assess for DSM-5 autism criteria.
  Eyelink Portable Duo: Eye movements and pupil diameter will be collected while participants view a series of developmentally appropriate pictures and movies. Children will be asked to sit in highchair or on a caregiver's lap and will face a computer monitor. The eye tracking portion of the visit will last approximately 15 minutes or until the child is no longer able to attend to pictures/videos.
  Integrated PCP Diagnosis and Eye-tracking Biomarker: A Classification and Regression Tree (CART) Analysis, based on recursive partitioning, was used to determine which combination of variables (EE Hub PCP diagnosis, diagnostic certainty, composite biomarker, and biomarker frequency [sum of all individual biomarkers (0-6) that exceeded the 95% specificity threshold for each child]) best predicted reference standard autism diagnosis.
Arm/Group | Children Undergoing Developmental Evaluation
Number analyzed (Participants) | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.55 (0.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 104
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race / ethnicity: Asian | 2
  Race / ethnicity: Black | 14
  Race / ethnicity: Latine, any race | 21
  Race / ethnicity: Non-Latine White | 96
  Race / ethnicity: More than one race | 6
  Race / ethnicity: Unspecified or not reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 146
Composite Eye-tracking Biomarker [Count of Participants; unit: Participants] — Participants with a composite eye-tracking biomarker indicative of autism
  Participants | 89

OUTCOME MEASURES:

1. Primary Outcome: Agreement Between Composite Eye-tracking Biomarker and Expert Autism-specialist
Description: Sensitivity and specificity of a composite eye-tracking (i.e., index) test, which was a consolidated measure based on significant eye-tracking indices, compared to reference standard expert clinical autism diagnosis.
Time Frame: Day 1
Population: The number of participants analyzed does not differ from the number of participants assigned to this arm.
Measure: Count of Participants; unit: Participants
Groups:
- Autism (Reference Standard): Reference standard autism diagnosis made by a licensed clinical psychologist with expertise in autism diagnosis based upon a research evaluation including the Autism Diagnostic Observation Schedule, Second Edition (ADOS-2), Vineland Adaptive Behaviors Scale, Third Edition (VABS-3), Mullen Scales of Early Learning (MSEL), and a caregiver interview to assess for DSM-5 autism criteria
- Non-Autism (Reference Standard): Reference standard non-autism diagnosis made by a licensed clinical psychologist with expertise in autism diagnosis based upon a research evaluation including the Autism Diagnostic Observation Schedule, Second Edition (ADOS-2), Vineland Adaptive Behaviors Scale, Third Edition (VABS-3), Mullen Scales of Early Learning (MSEL), and a caregiver interview to assess for DSM-5 autism criteria
Arm/Group | Autism (Reference Standard) | Non-Autism (Reference Standard)
Number analyzed (Participants) | 102 | 44
Participants
  Autism (index test) | 79 | 10
  Non-autism (index test) | 23 | 34

2. Primary Outcome: Agreement Between Integrated PCP, Eye-tracking Biomarker Score and Expert Autism-specialist
Description: Classification and Regression Tree (CART) analysis, based on recursive partitioning, is used to determine which combination of variables (EE Hub PCP diagnosis, diagnostic certainty, composite biomarker, and biomarker frequency [sum of all individual biomarkers (0-6) that exceeded the 95% specificity threshold for each child]) best predicted reference standard autism diagnosis.
Time Frame: Day 1
Population: Because the goal of tiered diagnostic models, such as the EAE Hub system, is that PCPs can rule in/out autism in a subset of children and refer more complicated cases to a specialist, terminal nodes for the CART analysis were identified as autism, non-autism, or refer. As such, the number of participants analyzed differs from the number of participants assigned to the arm. A total of 19 children were classified as refer, and thus the total number of participants was 127.
Measure: Count of Participants; unit: Participants
Arm/Group | Autism (Reference Standard) | Non-Autism (Reference Standard)
Number analyzed (Participants) | 97 | 30
Participants
  Autism (index text) | 88 | 4
  Non-Autism (index text) | 9 | 26

ADVERSE EVENTS:
Time Frame: 1 Day
Arm/Group | Children Undergoing Developmental Evaluation
All-Cause Mortality (participants affected / at risk) | 0/154
Serious Adverse Events (participants affected / at risk) | 0/154
Other Adverse Events (participants affected / at risk) | 0/154

LIMITATIONS AND CAVEATS:
While the current study included a prospective, consecutively-referred sample of children evaluated for autism, a class imbalance was present; such an imbalance has the potential to overinflate accuracy metrics, and thus our findings should be interpreted with caution. Although 95% of children provided at least one usable eye-tracking measure, the percentage of usable data across each task varied significantly (50-94%).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/88/NCT06586788/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/88/NCT06586788/ICF_001.pdf